CLINICAL TRIAL: NCT02844647
Title: Hyperpolarized Carbon-13 Imaging of Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 432-2015
Record Dates: First submitted 2016-06-13; First posted 2016-07-26 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI w/ Hyperpolarized Pyruvate (13C) (Experimental): "Hyperpolarization" of low natural abundance species such as 13C, when injected offers the potential of extracting metabolic information by real-time MR imaging of biochemical reactions within the body. The biochemical reactions, including lactate production, will be measured using MRI.
  Interventions: Other: Hyperpolarized Pyruvate (13C)

INTERVENTIONS:
Other: Hyperpolarized Pyruvate (13C) — MRI contrast agent

SUMMARY:
A pilot study with a group of up to 10 men with CRPC about to embark on a 6-month course of treatment with radium 223. Study participants will undergo anatomical MR imaging combined with the new hyperpolarized MRI (1 hour exam) prior to treatment.

DETAILED DESCRIPTION:
"Hyperpolarization" of low natural abundance species such as 13C, offers the potential of extracting metabolic information by real-time imaging of biochemical reactions within the body. In this project, the investigators focus on prostate cancer, specifically late-stage disease, as management of these patients would benefit from a new imaging method that enables improved therapy selection, planning and monitoring.

For imaging the lactate distribution in bone-metastatic prostate cancer, 3D coverage of a large field-of-view is required in order to cover the vertebral column (the most common site of metastases). To enable this, the investigators have developed methods using a large-volume transmitter and multi-channel receiver system for 3-dimensional 13C metabolic imaging in these patients. The image resolution and encoding matrix were tailored to the required 3D coverage of the vertebral column.

At the end of this study, the investigators will have the methodology, hardware and clinical-research workflow needed to evaluate 13C-lactate imaging as a new tool to help patients with metastatic prostate cancer. The investigators would be the first in the world to apply 13C metabolic MRI to bone metastases. Although the investigators propose to study patients who are starting a 6-month course of treatment with radium 223, in this project, this proof-of-concept study may also lead to a larger clinical trial at different points in the treatment pathway, such as prior to deciding between treatment with cytotoxic agents versus drugs that target the androgen axis such as abiraterone.

ELIGIBILITY:
Inclusion Criteria:

* Men with bone-metastatic CRPC before starting the first dose of radium 223 therapy
* Laboratory requirements:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x109/L
* Hemoglobin ≥ 10.0 g/dL (100 g/L; 6.2 mmol/L)
* Total bilirubin level ≤ 1.5 institutional upper limit of normal (ULN)
* ASAT and ALAT ≤ 2.5 ULN
* • Creatinine ≤ 1.5 ULN
* Albumin >25 g/L
* Eastern Cooperative Oncology Group Status of 0 or 1

Exclusion Criteria:

* Unable to give valid informed consent
* Contraindication for MRI as per Sunnybrook MRI questionnaire (Appendix 1).
* Claustrophobia
* Body mass index of less than 18.5 or greater than 32
* Congestive heart failure, a past or present medical history of clinically significant electrocardiogram (EKG) abnormalities, which may include QT prolongation, a family history of prolonged QT interval syndrome, or a myocardial infarction (MI) within the past 12 months with ensuing unstable EKG, or ongoing acute or chronic pulmonary bronchospastic disease, including a history of chronic obstructive pulmonary disease or asthma, with an exacerbation within the past year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Images of lactate, bicarbonate and pyruvate in patients with bone-metastatic CRPC measured by MRI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cunningham, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No